CLINICAL TRIAL: NCT02839746
Title: Non-interventional Study Describing Treatment Convenience in Patients Treated With Dabigatran for Stroke Prophylaxis in Atrial Fibrillation (SPAF)
Brief Title: Treatment Convenience in Patients Treated With Dabigatran for Stroke Prophylaxis in Atrial Fibrillation (SPAF)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.253
Record Dates: First submitted 2016-06-02; First posted 2016-07-21 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Dabigatran: Patients switched from vitamin K antagonist (VKA) to dabigatran

SUMMARY:
Describe patient and physician assessed factors for patient well-being when treated with Pradaxa for stroke and embolism prevention in atrial fibrillation either compared to previous antithrombotic treatment (switcher)

ELIGIBILITY:
Inclusion criteria:

* Written informed consent prior to participation
* Female and male patients 18 years of age or older with a diagnosis of non-valvular atrial fibrillation.
* At least 6 months of continuous vitamin K antagonist (VKA) treatment for stroke prevention prior to baseline assessment.
* Patients switched to Pradaxa® according to Summary of Product Characteristics, therapeutic positioning report from Spanish competent authorities and visa from each autonomous community.

Exclusion criteria:

* Contraindication to the use of Pradaxa® or VKA as described in the Summary of Product Characteristics (SmPC)
* Patients receiving Pradaxa® or VKA for any other condition than stroke prevention in non-valvular atrial fibrillation.
* Current participation in any clinical trial of a drug or device

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: spanish patients with a diagnosis of non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data collection periods:
  * When planned to be switched from vitamin K antagonists (VKA) to Pradaxa® (At baseline, Visit 1)
  * 7 to 124 days after starting treatment with Pradaxa® (initiation period, Visit 2)
  * 125 to 365 days after starting treatment with Pradaxa® (continuation period, Visit 3)
  Questionnaire (quest.)
Pre-assignment Details: All participants were screened for eligibility to participate in the study. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered if any one of the specific entry criteria were not met.
Groups:
- Dabigatran Etexilate (Pradaxa®): Patients with Non-valvular atrial fibrillation (NVAF) who were treated with vitamin K antagonists (VKAs) and subsequently started daily oral dose of Pradaxa® 110 milligram (mg) or 150 mg hard capsules containing dabigatran etexilate according to the Summary of Product characteristics, therapeutic positioning report from Spanish competent authorities and visa from each autonomous community.
Period: Overall Study
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Started | 671
Completed | 659
Not Completed | 12
Not completed — Not met selection criteria | 12

BASELINE CHARACTERISTICS:
Population: Eligible patients: All patients (pts) fulfilling all inclusion criteria and no exclusion criteria.
Groups:
- Total: Patients with Non-valvular atrial fibrillation (NVAF) who were treated with vitamin K antagonists (VKAs) and subsequently started daily dose of Pradaxa® 110 mg or 150 mg hard capsules containing dabigatran etexilate according to the Summary of Product characteristics, therapeutic positioning report from Spanish competent authorities and visa from each autonomous community.
Arm/Group | Total
Number analyzed (Participants) | 659
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.12 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275
  Male | 384
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race information is provided. Ethnicity information was not collected for this study.
  Participants
    Caucasian | 638
    North African | 2
    Latin American | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean of Perception of Anticoagulant Treatment Questionnaire 2 (PACT-Q2) Scores at Second Assessment Compared to Baseline Assessment
Description: The PACT-Q is self-administered quest. which was developed as means to investigate patients' satisfaction with anticoagulant treatment & treatment convenience in patients with deep venous thrombosis (DVT), pulmonary embolism (PE) or atrial fibrillation (AF). PACT-Q2 quest. is made up of two domains: (1) Convenience (13 items): This domain is calculated by adding inverted scores (6-item score) for each of the 13 items in question & converting to a scale from 0 to 100. (2) Satisfaction with the anticoagulant treatment (7 items): This domain is calculated by adding scores for each of the 7 items in question & converting to a scale from 0 to 100. The missing items have been replaced by the mean of non-missing items of the dimension (if 50% of items were completed, non-missing), in order to calculate domains score. The higher the score, the higher the convenience/satisfaction. The two domain scores are presented for Baseline, Visit 2 (second assessment) as mean & standard deviation (SD).
Time Frame: When planned to be switched from VKA to Pradaxa® (At baseline, Visit 1), 7 to 124 days after starting treatment with Pradaxa® (initiation period, Visit 2)
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria. The analyses were performed based on actual anticoagulant treatment (AT) received by pts (i.e. "as-treated" analysis),so that pts who discontinued the initial AT during time of an assessment were excluded from all analyses where data from that assessment was included
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Units on Scale
  Convenience-Baseline: number analyzed (Participants) | 512
  Convenience-Baseline | 59.86 (25.39)
  Convenience-Visit 2: number analyzed (Participants) | 512
  Convenience-Visit 2 | 80.96 (16.98)
  Satisfaction-Baseline: number analyzed (Participants) | 511
  Satisfaction-Baseline | 49.15 (17.88)
  Satisfaction-Visit 2: number analyzed (Participants) | 511
  Satisfaction-Visit 2 | 69.35 (14.26)
Statistical Analysis 1: Comparison: Dabigatran Etexilate (Pradaxa®); Within group comparison of Baseline convenience with that of Visit 2; Test type: Other; p < 0.0001, non-parametric Wilcoxon signed-rank
Statistical Analysis 2: Comparison: Dabigatran Etexilate (Pradaxa®); Within group comparison of Baseline satisfaction with that of Visit 2; Test type: Other; p < 0.0001, non-parametric Wilcoxon signed-rank

2. Primary Outcome: Mean of Perception of Anticoagulant Treatment Questionnaire 2 (PACT-Q2) Scores at Last Assessment Compared to Baseline Assessment
Description: The PACT-Q is self-administered quest. which was developed as means to investigate patients satisfaction with anticoagulant treatment & treatment convenience in patients with deep venous thrombosis (DVT), pulmonary embolism (PE) or atrial fibrillation (AF). The PACT-Q2 quest. is made up of two domains: 1) Convenience (13 items): This domain is calculated by adding inverted scores (6-item score) for each of the 13 items in question, &converting to a scale from 0 to 100. 2) Satisfaction with the anticoagulant treatment (7 items):This domain is calculated by adding scores for each of the 7 items in question, & converting to a scale from 0 to 100.
  The missing items have been replaced by the mean of non-missing items of the dimension (if 50% of items were completed, non-missing), in order to calculate domains score. The higher the score, the higher the convenience/satisfaction.
  The two domain scores are presented for Baseline, Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: When planned to be switched from VKA to Pradaxa® (At baseline, Visit 1), 125 to 365 days after starting treatment with Pradaxa® (continuation period, Visit 3)
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.The analyses were performed based on actual anticoagulant treatment (AT) received by pts (i.e. "as-treated" analysis),so that pts who discontinued the initial AT during time of an assessment were excluded from all analyses where data from that assessment was included
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Units on Scale
  Convenience-Baseline: number analyzed (Participants) | 491
  Convenience-Baseline | 60.19 (25.59)
  Convenience-Visit 3: number analyzed (Participants) | 491
  Convenience-Visit 3 | 84.29 (15.19)
  Satisfaction-Baseline: number analyzed (Participants) | 489
  Satisfaction-Baseline | 49.44 (17.74)
  Satisfaction-Visit 3: number analyzed (Participants) | 489
  Satisfaction-Visit 3 | 73.19 (14.80)
Statistical Analysis 1: Comparison: Dabigatran Etexilate (Pradaxa®); Within group comparison of Baseline convenience with that of Visit 3; Test type: Other; p < 0.0001, non-parametric Wilcoxon signed-rank
Statistical Analysis 2: Comparison: Dabigatran Etexilate (Pradaxa®); Test type: Other — Within group comparison of Baseline satisfaction with that of Visit 3; p < 0.0001, non-parametric Wilcoxon signed-rank]

3. Primary Outcome: Mean of Perception of Anticoagulant Treatment Questionnaire (PACT-Q2) Score at Last Assessment Compared to Second Assessment
Description: The PACT-Q is self-administered quest. which was developed as means to investigate patients satisfaction with anticoagulant treatment & treatment convenience in patients with DVT, PE or AF. The PACT-Q2 quest. is made up of two domains: 1) Convenience (13 items): This domain is calculated by adding inverted scores (6-item score) for each of the 13 items in question, &converting to a scale from 0 to 100. 2) Satisfaction with the anticoagulant treatment (7 items):This domain is calculated by adding scores for each of the 7 items in question, & converting to a scale from 0 to 100. The missing items have been replaced by the mean of non-missing items of dimension (if 50% of items were completed, non-missing), in order to calculate domains score. The higher the score, the higher the convenience/satisfaction.
  The two domain scores are presented for Visit 2( second assessment), Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: 7 to 124 days after starting treatment with Pradaxa® (initiation period, Visit 2), 125 to 365 days after starting treatment with Pradaxa® (continuation period, Visit 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
unit on scale
  Convenience-Visit 2: number analyzed (Participants) | 486
  Convenience-Visit 2 | 80.95 (17.01)
  Convenience-Visit 3: number analyzed (Participants) | 486
  Convenience-Visit 3 | 84.23 (15.24)
  Satisfaction-Visit 2: number analyzed (Participants) | 483
  Satisfaction-Visit 2 | 69.54 (14.22)
  Satisfaction-Visit 3: number analyzed (Participants) | 483
  Satisfaction-Visit 3 | 73.30 (14.66)
Statistical Analysis 1: Comparison: Dabigatran Etexilate (Pradaxa®); Within group comparison of visit 2 convenience with that of Visit 3; Test type: Other; p < 0.0001, non-parametric Wilcoxon signed-rank
Statistical Analysis 2: Comparison: Dabigatran Etexilate (Pradaxa®); Within group comparison of visit 2 satisfaction with that of Visit 3; Test type: Other; p < 0.0001, non-parametric Wilcoxon signed-rank

4. Secondary Outcome: Patient Characteristics at Baseline - CHA2DS2-VASc Stroke Risk Score and HAS-BLED Bleeding Risk Score
Description: CHA2DS2-VASc stroke risk score is calculated based on following conditions: Congestive heart failure/left ventricular dysfunction, Hypertension, Age (≥ 75), Diabetes Mellitus,Stroke/Transient Ischaemic Attack (TIA)/thromboembolism,Vascular disease (history of myocardial infarction, peripheral artery disease or aortic plaque) ,Age 65-74, Sex category. HAS-BLED bleeding risk score is calculated based on following conditions: Uncontrolled hypertension with Systolic Blood pressure (SBP) ≥ 160 mmHg,Kidney failure,liver failure,History of stroke,History of bleeding, anaemia or predisposition to bleeding,Unstable/high or poor international normalized ratio (INR) (<60% of time within therapeutic range),Elderly (>65 years),Medications that affect haemostasis,Consumptions of ≥8 alcoholic drinks per week.CHA2DS2-VASc stroke risk score & HAS-BLED bleeding risk score range from 0 to 9 with 0 being outcome with low stroke risk for CHA2DS2-VASc and being with low bleeding risk for HAS-BLED.
Time Frame: Baseline
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
unit on scale
  CHA2DS2-VASc | 3.60 (1.56)
  HAS-BLED | 2.10 (0.98)

5. Secondary Outcome: Patient Characteristics at Baseline - Categorical Parameters
Description: Categorical parameters of the patient characteristics at baseline included age, Risk factors associated with stroke and/or haemorrhage in the medical history (MH), co-morbidities (CoMo), concomitant medication (CM) and dosing of Pradaxa® (DoP).
  Haemorrhagic risk (HAS-BLED) is categorized as Low risk (score 0), Moderate risk (score 1-2) and High Risk (score ≥3). Thromboembolic risk (CHA2DS2-VASc) is categorized as Low risk (score 0 in male and 1 in female), Moderate risk (score 1 in male and 2 in female) and High Risk (score ≥2 in male and ≥3 in female).
  Stages of kidney disease are categorized based on Cockcroft-Gault review as below:
  No kidney failure (> 80 ml/min), Mild kidney failure (50-80 ml/min), Moderate kidney failure (30-49 ml/min), Severe kidney failure (15-29 ml/min) and End-stage kidney failure/dialysis (< 15 ml/min).
Time Frame: Baseline
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Participants
  Age: ≤65 years | 132
  Age: >65 years | 527
  MH: Ischaemic stroke | 88
  MH: Thromboembolisms | 17
  MH: Diabetes mellitus | 159
  MH: Arterial hypertension | 351
  MH: Ischemic heart disease or Heart failure | 136
  MH: Peripheral arterial disease | 19
  MH: Kidney failure | 9
  MH: Liver failure | 5
  CoMo: Yes | 425
  CoMo: No | 231
  CoMo: Not assessed | 3
  CM: Yes | 597
  CM: No | 62
  DoP: 110 mg twice daily | 244
  DoP: 150 mg twice daily | 415
  HAS-BLED: Low | 23
  HAS-BLED: Moderate | 435
  HAS-BLED: High | 201
  CHA2DS2-VASc: Low | 8
  CHA2DS2-VASc: Moderate | 60
  CHA2DS2-VASc: High | 591
  No kidney failure: number analyzed (Participants) | 643
  No kidney failure | 211
  Mild kidney failure: number analyzed (Participants) | 643
  Mild kidney failure | 385
  Moderate kidney failure: number analyzed (Participants) | 643
  Moderate kidney failure | 44
  Severe kidney failure: number analyzed (Participants) | 643
  Severe kidney failure | 3
  End-stage kidney failure/dialysis: number analyzed (Participants) | 643
  End-stage kidney failure/dialysis | 0

6. Secondary Outcome: Patient Characteristics at Baseline - Creatinine Clearance
Description: Creatinine clearance at baseline is a measure of the patient's kidney function and is one of the baseline patient characteristics.
Time Frame: Baseline
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Mean (Standard Deviation); unit: millilitre/ minute [mL/min]
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
millilitre/ minute [mL/min] | 73.91 (22.72)

7. Secondary Outcome: Patient Characteristics at Baseline - Vitamin K Antagonist Treatment Duration
Description: Vitamin K Antagonist (VKA) treatment duration is one of the baseline patient characteristics.
Time Frame: Baseline
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Months | 47.83 (46.51)

8. Secondary Outcome: Patient Characteristics at Baseline - Reasons for Switching From VKAs to Pradaxa®
Description: Categories of reasons for switching from VKAs to Pradaxa® are as below:
  1. Hypersensitivity (Hypersensitivity to the drug)
  2. Intracranial haemorrhage (Patients with a history of intracranial haemorrhage (ICH) (except during the acute phase) in whom the benefits of anticoagulation were deemed to outweigh the risk of haemorrhage)
  3. Ischaemic stroke (Patients with ischaemic stroke who present clinical and neuroimaging criteria indicating a high risk of ICH)
  4. Arterial thromboembolic episodes (Patients undergoing treatment with VKAs, suffering from severe arterial thromboembolic episodes despite good INR control)
  5. INR not in range (Patients who have started treatment with VKAs in whom it is not possible to keep the INR in range (2-3) despite good therapeutic compliance)
  6. INR management (Lack of access to conventional INR management)
  7. Pts decision (Patient's decision)
  8. Others.
  A single patient may have specified more than one reason
Time Frame: Baseline
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Participants
  Hypersenstitivity | 6
  Intracranial haemorrhage | 6
  Ischaemic stroke | 14
  Arterial thromboembolic episodes | 29
  INR not in range | 484
  INR management | 45
  Pts decision | 137
  Other | 13

9. Secondary Outcome: Reason for Changing the Dose of Pradaxa®: 150 mg/ Twice Daily (Bid) to 110 mg/Bid
Description: Reasons for for changing the dose of Pradaxa®: 150 mg/bid to 110 mg/bid are categorized as below:
  1] High risk of bleeding 2] Moderate renal failure 3] >80 years 4] Other reason
Time Frame: as for outcome 3
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Participants
  High risk of bleeding- Visit 2: number analyzed (Participants) | 620
  High risk of bleeding- Visit 2 | 2
  Moderate renal failure- Visit 2: number analyzed (Participants) | 620
  Moderate renal failure- Visit 2 | 1
  >80 years- Visit 2: number analyzed (Participants) | 620
  >80 years- Visit 2 | 0
  Other reason- Visit 2: number analyzed (Participants) | 620
  Other reason- Visit 2 | 2
  High risk of bleeding- Visit 3: number analyzed (Participants) | 586
  High risk of bleeding- Visit 3 | 0
  Moderate renal failure- Visit 3: number analyzed (Participants) | 586
  Moderate renal failure- Visit 3 | 3
  >80 years- Visit 3: number analyzed (Participants) | 586
  >80 years- Visit 3 | 2
  Other reason- Visit 3: number analyzed (Participants) | 586
  Other reason- Visit 3 | 2

10. Secondary Outcome: Reason for Changing the Dose of Pradaxa®: 110 mg/Bid to 150 mg/Bid
Description: Reasons for for changing the dose of Pradaxa®: 110 mg/bid to 150 mg/bid are categorized as below:
  1] High risk of bleeding 2] Moderate renal failure 3] >80 years 4] Other reason
Time Frame: as for outcome 3
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Participants
  High risk of bleeding- Visit 2: number analyzed (Participants) | 620
  High risk of bleeding- Visit 2 | 0
  Moderate renal failure- Visit 2: number analyzed (Participants) | 620
  Moderate renal failure- Visit 2 | 0
  >80 years- Visit 2: number analyzed (Participants) | 620
  >80 years- Visit 2 | 0
  Other reason- Visit 2: number analyzed (Participants) | 620
  Other reason- Visit 2 | 1
  High risk of bleeding- Visit 3: number analyzed (Participants) | 586
  High risk of bleeding- Visit 3 | 0
  Moderate renal failure- Visit 3: number analyzed (Participants) | 586
  Moderate renal failure- Visit 3 | 0
  >80 years- Visit 3: number analyzed (Participants) | 586
  >80 years- Visit 3 | 0
  Other reason- Visit 3: number analyzed (Participants) | 586
  Other reason- Visit 3 | 2

11. Secondary Outcome: Reasons for no Longer Receiving Pradaxa® Treatment
Description: Reasons for no longer receiving Pradaxa® treatment categorized as below:
  1. Treatment change (Change of treatment (by patient or by investigator)
  2. Adverse event (Diarrhea, gastrointestinal discomfort, rectorrhagia, dyspepsia)
  3. Exitus
  4. Others
Time Frame: as for outcome 3
Population: Eligible pts: All pts fulfilling all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 659
Participants
  Treatment change- Visit 2: number analyzed (Participants) | 26
  Treatment change- Visit 2 | 8
  Adverse event- Visit 2: number analyzed (Participants) | 26
  Adverse event- Visit 2 | 10
  Exitus- Visit 2: number analyzed (Participants) | 26
  Exitus- Visit 2 | 1
  Other reason- Visit 2: number analyzed (Participants) | 26
  Other reason- Visit 2 | 7
  Treatment change- Visit 3: number analyzed (Participants) | 27
  Treatment change- Visit 3 | 7
  Adverse event-- Visit 3: number analyzed (Participants) | 27
  Adverse event-- Visit 3 | 7
  Exitus- Visit 3: number analyzed (Participants) | 27
  Exitus- Visit 3 | 6
  Other reason- Visit 3: number analyzed (Participants) | 27
  Other reason- Visit 3 | 7

ADVERSE EVENTS:
Time Frame: From signing the informed consent till end of the study; up to 365 days
Arm/Group | Dabigatran Etexilate (Pradaxa®)
All-Cause Mortality (participants affected / at risk) | 8/653
Serious Adverse Events (participants affected / at risk) | 14/653
Other Adverse Events (participants affected / at risk) | 0/653
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Pradaxa®) (N=653)
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Influenza (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT02839746/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT02839746/SAP_001.pdf